CLINICAL TRIAL: NCT07222085
Title: Determining the Long-Term Stability of the Glide Control Strategy for Upper Limb Prostheses
Brief Title: Long-Term Stability of the Glide Control Strategy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Infinite Biomedical Technologies (Industry)
Collaborators: Medical Center Orthotics and Prosthetics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OR240247
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Upper Limb Amputation Above Elbow; Upper Limb Amputation Below Elbow
Keywords: Glide; Pattern Recognition; Myoelectric Control; Upper Limb Prostheses

STUDY DESIGN:
Intervention Model Description: The study participants will then be randomly block assigned to one of two groups in pair: Group AB will be prescribed a commercial Pattern Recognition (PR) system for the first Phase of the take-home evaluation and Glide for the second Phase. Group BA will be prescribed the control strategies in the inverse order, using Glide during the first Phase and a commercial PR system during the second. Within each group, participants will be again randomly assigned into one of three subgroups: AB10, AB12, and AB14 (or BA10, BA12, and BA14). These subgroups determine the duration of the first (i.e., baseline) Phase, with subgroups correlating to 10-weeks, 12-weeks, and 14-weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Glide then Pattern Recognition (Experimental): Participants use a Glide-controlled upper limb prosthesis first, followed by a Pattern Recognition-based upper limb prosthesis.
  Interventions: Device: Glide Control System; Device: Pattern Recognition System
- Pattern Recognition then Glide (Experimental): Participants use a Pattern Recognition-based upper limb prosthesis first, followed by a Glide-controlled upper limb prosthesis.
  Interventions: Device: Glide Control System; Device: Pattern Recognition System

INTERVENTIONS:
Device: Glide Control System — Glide is a commercially developed directional myoelectric control strategy from Infinite Biomedical Technologies (IBT) that sits between classic Direct Control (DC) and modern Pattern Recognition (PR). Instead of requiring an isolated on/off muscle signal for each function (e.g., DC) or training a complex classifier on many gestures (e.g., PR), Glide uses the relative activity across 2-8 EMG electrodes to move a virtual cursor on a 2-D "Glide map." The map is divided into adjustable sectors ("slices"), and each slice is assigned a prosthetic movement (e.g., hand open/close, wrist rotation, elbow flexion). Moving the cursor into a slice actuates that movement.
Device: Pattern Recognition System — Pattern recognition (PR)-based myoelectric control is a data-driven approach that allows a user to control multiple prosthetic functions using natural muscle activation patterns rather than discrete, isolated signals. Instead of mapping one muscle to one motion (as in conventional Direct Control), PR systems record the spatial and temporal pattern of EMG activity from multiple sites on the residual limb and use machine learning algorithms to classify which intended movement the user is trying to make.

SUMMARY:
This research is intended to test whether the prescription of the Glide prosthesis control system reduces the burden of use for both patients and their clinical care team as compared to use of Pattern Recognition-based advanced myoelectric control. The goal of the study is to fill the gaps in clinically relevant knowledge to inform the prescription of prosthesis components and the rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral trans-radial or trans-humeral limb loss with a healed residual limb
* Candidate for 2+ degree-of-freedom (DOF) myoelectric prosthesis as determined by the study prosthetist
* Age of 18 years or greater

Exclusion Criteria:

* Prior experience with Pattern Recognition or Glide control
* Individuals with a residual limb that is unhealed from the amputation surgery
* Individuals with easily damaged or sensitive skin who would not tolerate EMG electrodes
* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon clinical evaluation
* Serious uncontrolled medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Daily Mean Number of Control Adjustment Sessions (DMNCAS) | Weekly, From Prosthesis Delivery (Day 0) to the End of Treatment (Day 168)
  DMNCAS quantifies the number of times a prosthesis user needs to adjust their control strategy to maintain performance. For a PR system, a control adjustment refers to a calibration (or recalibration) of one or more prosthesis movements, while for the Glide control strategy, a control adjustment refers to a change in the Glide map configuration (e.g., electrode gains, slice geometries, assigned movements, etc.). A control adjustment session is then a period of time devoted to performing one or more control adjustments. The number and duration of control adjustment sessions will be recorded in a study diary.
Number of Follow-Up Clinical Interventions (NFCI) | Weekly, From Prosthesis Delivery (Day 0) to End of Treatment (Day 168)
  NFCI reports the number of times the prosthesis user requests the aid of a clinician to resolve an issue with their prescribed control strategy. NFCI refers to clinical interventions (both remote and in-person) that occur post-prosthesis delivery, the number and duration of which will be recorded in a study diary. Diary entries will be verified through a retrospective chart review in collaboration with Medical Center Orthotics & Prosthetics.

SECONDARY OUTCOMES:
Socket Comfort Score (SCS) | Weekly, From Prosthesis Delivery (Day 0) to End of Treatment (Day 168)
  SCS is a validated, 11-point numerical rating scale that quantifies a respondent's subjective experience of comfort while wearing a prosthesis. The score ranges from 0 (or "the least comfortable socket fit you can imagine") to 10 (or "the most comfortable socket you can imagine"). A higher score indicates a more comfortable socket fit. Full administration of the SCS is estimated to take about 5 minutes.
Numerical Pain Rating Scale (NPRS) | Weekly, From Prosthesis Delivery (Day 0) to End of Treatment (Day 168)
  NPRS is a pain screening tool that uses two 0 to 10 scales to measure pain intensity over the last seven days. The two scales interrogate different dimensions of pain: 1) residual limb pain; and 2) phantom limb pain. Both scales include descriptive anchors at the extremes (i.e., "no pain" is 0 and "the highest pain you can imagine" is 10). A higher score indicates a more intense pain experience. Full administration of the NPRS is estimated to take about 5 minutes.
PROMIS Pain Interference - Short Form 4a | Weekly, From Prosthesis Delivery (Day 0) to End of Treatment (Day 168)
  PROMIS Pain Interference short form 4a is a validated, self-report questionnaire that assesses consequences of pain on relevant aspects of one's life, including the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. The assessment comprises of four, 5-point Likert-type questions, each querying the respondent on their experience of pain in the previous seven days. PROMIS instruments are scored on a T-score metric (0 - 100) in which 50 is the mean of the reference population and 10 is the standard deviation. In general, a higher score equals more of the concept being measured. For the PROMIS Pain Interference questionnaire, a higher score then indicates a greater degree to which individuals believe pain interferes with their daily lives. Full administration of the PROMIS Pain Interference short form 4a is estimated to take about 5 minutes.
PROMIS Satisfaction - Short Form 8a | Weekly, From Prosthesis Delivery (Day 0) to End of Treatment (Day 168)
  PROMIS Satisfaction short form 8a is a validated, self-report questionnaire designed to query individuals on their satisfaction with their ability to participate in social roles and activities. The survey consists of eight, 5-point Likert-type questions covering several aspects of social engagement, including work, recreation, and maintaining interpersonal relationships. A higher score indicates a higher satisfaction with the respondent's ability to participate in work and home life. Full administration of the PROMIS Satisfaction short form 8a is estimated to take about 10 minutes.
OPUS Upper Extremity Functional Scale (UEFS) | Weekly, From Prosthesis Delivery (Day 0) to End of Treatment (Day 168)
  OPUS UEFS is a validated, self-report questionnaire that asks respondents to score how easily they can complete several activities of daily living (e.g., drink from a paper cup, brush hair, etc.). It is a low burden measure that provides a subjective view of a participant's functionality with a prosthesis. OPUS UEFS includes a total of 28 questions, each regarding an activity of daily living. Responses are divided into two parts: 1) a 5-point, Likert-type scale with descriptive anchors for each Level of Ease (e.g., "Cannot perform activity" is 0, "Very easy" is 4); and 2) an indication on if the activity is usually performed with or without a prosthesis. Participants may also provide a null response (i.e., "Not applicable") if they believe that the activity does not apply to them. The total score of the OPUS UEFS is the sum of the 28 responses converted to a Rasch measure (0 - 100). Higher scores therefore indicate greater functionality. Full administration takes about 25 minutes.
Mean Daily Prosthesis Wear Duration (MDPWD) | Weekly, From Prosthesis Delivery (Day 0) to End of Treatment (Day 168)
  MDPWD acts as a proxy for improved prosthesis acceptance. Prosthesis wear time is defined as the time from when participants don their prostheses to the time they doff their prostheses. Prosthesis wear duration is self-reported (in hours) by participants via a study diary.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Medical Center Orthotics and Prosthetics - Annapolis, Annapolis, Maryland
  - Medical Center Orthotics and Prosthetics - Baltimore, Baltimore, Maryland
  - Medical Center Orthotics and Prosthetics - Silver Spring, Silver Spring, Maryland
  - Medical Center Orthotics and Prosthetics - Allston, Allston, Massachusetts
  - Medical Center Orthotics and Prosthetics - Milton, Milton, Massachusetts
  - Medical Center Orthotics and Prosthetics - Charlotte, Charlotte, North Carolina
  - Medical Center Orthotics and Prosthetics - Anderson, Anderson, South Carolina
  - Medical Center Orthotics and Prosthetics - Greenville, Greenville, South Carolina
  - Medical Center Orthotics and Prosthetics - Fairfax, Fairfax, Virginia
  - Medical Center Orthotics and Prosthetics - Leesburg, Leesburg, Virginia